CLINICAL TRIAL: NCT00147368
Title: Pharmacokinetic-Pharmacodynamic Study of Adjunctive Arginine in Falciparum Malaria
Brief Title: Arginine Malaria Trial: Study of Adjunctive Arginine in Falciparum Malaria
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Wellcome Trust (Other); National Health and Medical Research Council, Australia (Other); MSHR (Unknown); National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other); Rumah Sakit Mitra Masyarakat Hospital (Other); University of Utah (Other); University of Sydney (Other)
Responsible Party: Nicholas Anstey, Menzies School of Health Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: arginine; GR071614MA - Wellcome Trust
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Malaria, Falciparum
Keywords: falciparum; malaria; arginine
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: intravenous (IV) arginine

SUMMARY:
Acute falciparum malaria is associated with low plasma arginine and impaired nitric oxide (NO) production. Both are associated with poor outcome. This study will examine the safety and effect of escalating doses of arginine in falciparum malaria. It will determine whether arginine can increase NO production and have an effect on NO-dependent physiological measurements. The hypothesis is that arginine: will be safe in falciparum malaria; will return plasma arginine concentration to normal/supranormal levels; will increase systemic and exhaled NO; reduces oxidant stress; and improves a number of NO-dependent physiological measures of relevance to malaria.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-60 years
2. P. falciparum parasitemia (1,000-100,000 parasites/ul).
3. Clinical syndrome consistent with malaria associated with documented fever (axillary temperature > 38℃) or self-reported history of fever in the last 48 hours with no other cause present
4. Commenced oral quinine ≤ 18 hours prior to scheduled commencement of arginine
5. An indication for hospital admission (eg relative cannot look after/supervise treatment at home but not having any warning signs or severe malaria criteria in "exclusion criteria" below)
6. Informed consent obtained

Exclusion Criteria:

1. Pregnancy or lactation
2. Mixed infection with P. falciparum and P. vivax
3. Warning signs of altered mental state and inability to sit unaided
4. Features of severe/complicated malaria
5. Diabetes
6. Systolic blood pressure (BP) < 100 mmHg
7. Serious underlying disease (cardiac, hepatic, kidney)
8. Initial iSTAT test showing any of the following values:

   * glucose < 4 mmol/L;
   * K+ ≥ 4.2 meq/L;
   * Cl- > 106 meq/L;
   * HCO3- < 20 meq/L.
9. Known allergy to L-arginine
10. Concurrent therapy with any of the following medications:

    * spironolactone;
    * oral nitrates;
    * phosphodiesterase inhibitor (eg sildenafil [Viagra]);
    * alpha-blocking antihypertensive agents (eg prazosin);
    * L-arginine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-02; Primary Completion 2006-04 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
exhaled and systemic nitric oxide production
endothelial function

SECONDARY OUTCOMES:
safety
pharmacokinetic (PK) parameters
pharmacodynamic (PD) parameters
oxidant stress
gas transfer
endothelial activation
a priori subgroup analysis: endothelial function in those with baseline impairment of function

CONTACTS AND LOCATIONS:
Overall Officials: Nick M Anstey, MBBS, Principal Investigator — MSHR
Locations (1):
- RSMM Hospital, Timika, Indonesia

REFERENCES:
- [Background] Yeo TW, Lampah DA, Gitawati R, Tjitra E, Kenangalem E, McNeil YR, Darcy CJ, Granger DL, Weinberg JB, Lopansri BK, Price RN, Duffull SB, Celermajer DS, Anstey NM. Impaired nitric oxide bioavailability and L-arginine reversible endothelial dysfunction in adults with falciparum malaria. J Exp Med. 2007 Oct 29;204(11):2693-704. doi: 10.1084/jem.20070819. Epub 2007 Oct 22. PMID 17954570
- [Derived] Yeo TW, Lampah DA, Gitawati R, Tjitra E, Kenangalem E, Granger DL, Weinberg JB, Lopansri BK, Price RN, Celermajer DS, Duffull SB, Anstey NM. Safety profile of L-arginine infusion in moderately severe falciparum malaria. PLoS One. 2008 Jun 11;3(6):e2347. doi: 10.1371/journal.pone.0002347. PMID 18545693